CLINICAL TRIAL: NCT02978235
Title: A Phase 1, Open-Label Safety, Pharmacokinetic and Efficacy Study of TAS4464 in Patients With Multiple Myeloma or Lymphoma
Brief Title: A Dose Finding Study Followed by a Safety and Efficacy Study for Patients With Multiple Myeloma or Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial was put on Clinical Hold and subsequently terminated prior to Phase 2 due to cases of drug induced liver injury meeting the criteria for Hy's Law
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAS-4464-101
Record Dates: First submitted 2016-11-21; First posted 2016-11-30 (Estimated); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Multiple Myeloma; NonHodgkin Lymphoma
Keywords: Multiple Myeloma; Relapsed/Refractory; Lymphoma; Non-Hodgkin Lymphoma; Diffuse Large B-Cell Lymphoma; DLBCL; Mantle Cell Lymphoma; MCL; Peripheral T-Cell Lymphoma; PTCL; TAS4464; NEDD8; NAE inhibitor; Neoplasms; Hematologic Diseases; Myeloma
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, Non-Hodgkin; Recurrence; Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Lymphoma, T-Cell, Peripheral; Neoplasms; Hematologic Diseases; Neoplasms, Plasma Cell | interventions — TAS4464

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TAS4464 (Experimental)
  Interventions: Drug: TAS4464

INTERVENTIONS:
Drug: TAS4464 — Intravenous (IV) Infusion

SUMMARY:
The Phase 1 portion of this study will determine the safety of TAS4464 and the most appropriate dose for patients with Multiple Myeloma or Lymphoma.

DETAILED DESCRIPTION:
The trial was put on Clinical Hold prior to Phase 2 due to cases of drug induced liver injury meeting the criteria for Hy's Law.

Background and Rationale:

• TAS4464 is an investigational NEDD8 activating enzyme (NAE) inhibitor, a compound which may affect cancer cell growth and survival. Thus, TAS4464 may help in the treatment of cancer.

Phase 1:

Primary:

* To investigate the safety and tolerability of TAS4464
* To identify a tolerated dose of TAS4464

Secondary:

* To investigate the preliminary efficacy of TAS4464
* To investigate the pharmacokinetics (PK) and the pharmacogenomics (PGx) of TAS4464
* To investigate the pharmacodynamics of TAS4464

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent
2. Women of child-bearing potential must have a negative pregnancy test

Multiple Myeloma:

Confirmed diagnosis of Multiple Myeloma with measurable disease, having been treated with at least two prior lines of therapy.

Lymphoma:

Confirmed diagnosis of Non-Hodgkin Lymphoma with measurable disease, having been treated with at least one anthracycline-based therapy, with relapse or progression since the last treatment received.

Exclusion Criteria:

1. Any of the following treatments, within the specified time frame, prior to the first dose of TAS4464:

   1. Major surgery within 28 days
   2. Radiation/chemotherapy within 21 days
   3. Monoclonal antibodies within 28 days
   4. Corticosteroid administration >20 mg/day of prednisone or equivalent within 14 days
   5. Proteasome inhibitors within 14 days
   6. Immunomodulatory agents within 7 days
   7. Stem cell transplant within 3 months
   8. Current immunosuppressive treatment for graft versus host disease
   9. Current use of an investigational agent
2. Active graft versus host disease
3. Known serious illness or medical condition
4. Prior treatment with TAS4464 or known hypersensitivity to any of its inactive ingredients or drugs similar in class
5. Pregnant or breast-feeding female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Number of patients experiencing any dose-limiting toxicities, during dose escalation period, to determine maximum tolerated dose of TAS4464, using NCI CTCAE criteria, laboratory testing, performance status assessments, and other routine visit procedures | Completion of Cycle 1 (28 days)
Efficacy of TAS4464, defined as Objective Response Rate (ORR) per IWG criteria (NHL) and IMWG criteria (MM). This will take into consideration routine assessments including: imaging scans, physical exams, blood tests, urine tests and biopsy results | Up to 5 years

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - John Theurer Cancer Center at Hackensack Meridian Health, Hackensack, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Gabrail Cancer Center, Canton, Ohio